CLINICAL TRIAL: NCT01430000
Title: Safety and Efficacy of Sustained Interferon Alfa 2b (INF) Therapy of Relapsing Hepatitis C (HCV) Patients Using InfraDure Biopump
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medgenics Medical Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG-002-01
Record Dates: First submitted 2011-09-04; First posted 2011-09-07 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Subcutan implantation of autologus skin graft after ex-vivo treatment — Subcutan implantation of autologus skin graft after ex-vivo treatment

SUMMARY:
Patients who completed the conventional treatment against HCV and relapsed (the virus appeared again in their blood) have no effective therapy.

DETAILED DESCRIPTION:
The rational behind the proposed study is that most patients can not tolerate the prolonged IFN injections because the side effects. The new proposed treatments allows continous low doses of IFN to be secreted by the patients himself using his own skin in which the dermo fibroblasts are enriched by a human gene of erythropoietin. The "biopump" continues to secret the IFN for several months avoiding the spikes of IFN in the plasma which are beleived to cause the undesired effects.

Patients will be able to complete a long treatment with low IFN dose and Ribavirin hoping to induce prolonged remission and cure

ELIGIBILITY:
Inclusion Criteria:

* Signed patient consent form
* Chronic HCV patients in relapse following conventional treatment regimen (INF+Ribavirine) with detectable plasma level of HCV RNA
* Hepatitis B and human immunodeficiency virus negative at screening visit
* Able and willing to follow contraception requirements
* Screening laboratory values, test, and physical exam within acceptable range

Exclusion Criteria:

* Current enrollment in another investigational device or drug study
* Anticipated inability to complete all clinic visits and comply with study procedures
* History of, or any current medical condition, which could impact the safety of the subject during the study
* Autoimmune hepatitis, suspected hepatocellular carcinoma, decompensated liver disease, or other known liver disease other than HCV
* Alcoholism or substance abuse with <6 documented months of sobriety
* Known allergy or sensitivity to interferons or ribavirin
* Any other condition that, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject participating in and completing the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy of Sustained Interferon Alfa 2b (INF) Therapy of Relapsing Hepatitis C (HCV) Patients using InfraDure Biopump | 9 months
  All subjects will receive autologous InfraDure Biopump tissue implants intended to provide sustained production and delivery of therapeutic levels of INF for up to three (3) months following INFRADURE Biopump implantation, with possibility of extension for an additional six months for a total of 9 month post INFRADURE Biopump implantation. Saftey parameters (Adverse events and Serious Adverse Events as well as immediate and long term tolerability are the main safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Eithan Galun, Professor, Principal Investigator — No affiliation
Locations (1):
- Prof. Eithan Galun Gene Therapy Institute, Hadassah Medical Center Ein Kerem, Jerusalem, Israel, Jerusalem, Jerusalem, Israel